CLINICAL TRIAL: NCT04156100
Title: A Phase 1 Study of AGEN1223, a Bispecific Fc-Engineered Antibody as a Single Agent and in Combination With Balstilimab, an Anti-PD-1 Monoclonal Antibody, in Subjects With Advanced Solid Tumors
Brief Title: A Study in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic business decision.
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-900-01
Record Dates: First submitted 2019-09-18; First posted 2019-11-07 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumor
Keywords: Cancer, Solid Tumor, PD-L1
MeSH Terms: conditions — Neoplasms | interventions — balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AGEN1223 (Experimental): AGEN1223 is a bispecific antibody.
  Interventions: Drug: AGEN1223
- AGEN1223 and balstilimab (Experimental): AGEN1223 is a bispecific antibody and balstilimab an anti-PD-1 Monoclonal Antibody
  Interventions: Drug: AGEN1223 and balstilimab

INTERVENTIONS:
Drug: AGEN1223 — AGEN1223 is a bispecific antibody.
  Arms: AGEN1223
Drug: AGEN1223 and balstilimab — AGEN1223 is a bispecific antibody and balstilimab an anti-PD-1 Monoclonal Antibody.
  Arms: AGEN1223 and balstilimab

SUMMARY:
This study is an open-label, Phase 1 study to evaluate the safety, tolerability, PK, and pharmacodynamic profiles of AGEN1223 as a single-agent and in combination with balstilimab, as well as to assess the maximum tolerated dose and determine the RP2D of AGEN1223 as a single-agent and in combination with balstilimab in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This study is an open-label, Phase 1 study to evaluate the safety, tolerability, PK, and pharmacodynamic profiles of AGEN1223 as a single-agent and in combination with balstilimab, as well as to assess the maximum tolerated dose and determine the RP2D of AGEN1223 as a single-agent and in combination with balstilimab in subjects with advanced solid tumors. This Phase 1 study will be conducted in an accelerated titration (for the first 2 single agent AGEN1223 dosing cohorts) and standard 3+3 dose escalation format. Study drug treatment will be administered on Day 1 of each 3-week cycle for up to 2 years or until any progressive disease (PD) or unacceptable toxicity is reported. The timing of the administration of doses may be adjusted for management of adverse events (AEs). The safe starting dose of AGEN1223 single-agent will be at the estimated minimally anticipated biological effect level.

The treatment phase is divided into 3-week cycles with associated evaluations and procedures that must be performed at specific time points. Tumor assessments will be conducted every 6 weeks (±7 days) from first dose until treatment discontinuation or disease progression. In subjects that discontinue treatment for reasons other than PD, imaging will continue until PD or initiation of a new therapy. If the subject discontinues treatment because of PD, imaging may be performed if clinically beneficial or if deemed necessary by the investigator until the initiation of new antineoplastic therapy. This must be approved by the Sponsor.

A Safety Monitoring Committee (SMC) will be established to assess safety and determine dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate by giving signed, dated, and written informed consent prior to any study specific procedures (participation in genetic testing is optional).
2. Greater than or equal to 18 years of age
3. Histologically or cytologically confirmed diagnosis of an advanced solid tumor for which no standard therapy is available or standard therapy has failed.
4. Measurable disease on baseline imaging based on RECIST 1.1.
5. Life expectancy of at least 3 months and an ECOG performance status of 0 or 1 (Appendix A).
6. Adequate organ function as indicated by the following laboratory values:

   * Adequate hematological function, defined as ANC ≥1.5 × 109/L, platelet count ≥100 × 109/L, and hemoglobin ≥8 g/dL without recent transfusion (defined as a transfusion that has occurred within 2 weeks of the hemoglobin measurement).
   * Adequate hepatic function based by a total bilirubin level ≤1.5 × the institutional upper limit of normal (IULN), AST level ≤2.5 × IULN, ALT level ≤2.5 × IULN.
   * Adequate renal function defined as creatinine ≤1.5 × IULN or measured or calculated creatinine clearance >40 mL/min per institutional standard. Assessment methods should be recorded.
   * Adequate coagulation defined by international normalized ratio or prothrombin time ≤1.5 × IULN and activated partial thromboplastin time ≤1.5 × IULN (unless the subject is receiving anticoagulant therapy).
7. No history of prior or concomitant malignancy that requires other active treatment.
8. Subjects must provide a sufficient and adequate FFPE tumor tissue sample (fresh biopsy) collected within 28 days before the first dose from a site not previously irradiated and to agree to a mandatory on-treatment biopsy if clinically feasible.
9. Female subjects of child-bearing potential must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication). Subjects with tumors producing human chorionic gonadotropin and gestational trophoblastic tumor do not need a serum pregnancy test, and absence of pregnancy should be documented by the Principal Investigator (PI) based on clinical and radiological assessments as needed. Non-childbearing potential is defined as:

   * ≥45 years of age and has not had menses for greater than 1 year,
   * Amenorrheic for ≥2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon prestudy (screening) evaluation,
   * Status is post-hysterectomy, oophorectomy, or tubal ligation.
10. Female subjects of child-bearing potential must be willing to use highly effective contraceptive measures starting with the screening visit through 90 days after the last dose of study treatment.

    Note: Abstinence is acceptable if this is the established and preferred contraception for the subject.
11. Male subjects with a female partner(s) of child-bearing potential must agree to use highly effective contraceptive measures throughout the study starting with the screening visit through 90 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

    Note: Abstinence is acceptable if this is the established and preferred contraception method for the subject.
12. Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 3 weeks of the first dose of current study drug.
2. Any relevant bispecific antibody, and/or anti-PD-1/PDL1 agents. For selected indication cohorts, prior treatment may be permitted after discussion with the Sponsor. Prior therapy with PD-1/PDL1 inhibitor may be allowed in agreement with the Sponsor.
3. Received prior systemic cytotoxic chemotherapy, biological therapy, radiotherapy, or major surgery within 3 weeks prior to first dose of study drug; a 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease with Sponsor approval.
4. Persisting toxicity with Grade >1 severity related to prior therapy based on NCI-CTCAE Version 5.0.

   Note: Sensory neuropathy and alopecia of Grade ≤2 are acceptable.
5. Expected to require any other form of systemic or localized antineoplastic therapy while on study (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
6. Known severe hypersensitivity reactions (NCI-CTCAE Grade ≥3) to fully human monoclonal antibodies, or severe reaction to immuno-oncology agents, such as colitis or pneumonitis, requiring treatment with steroids, or has a history of interstitial lung disease (ILD), any history of anaphylaxis, or uncontrolled asthma.
7. Receiving systemic corticosteroid therapy 1 week prior to the first dose of study drug or receiving any other form of systemic immunosuppressive medication.

   Note: Corticosteroid use as a premedication for IV contrast allergies/reactions is allowed. Subjects who are receiving daily corticosteroid replacement therapy are an exception to this rule. Daily prednisone at doses of up to 7.5 mg or equivalent hydrocortisone doses are examples of permitted replacement therapy. Use of inhaled or topical corticosteroids is permitted.
8. CNS tumor, metastasis, and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period or identified prior to consent.

   Note: Subjects with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions at screening (defined as 2 brain images, both of which are obtained after treatment to the brain metastases; these imaging scans should both be obtained ≥4 weeks apart). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have returned to baseline or resolved. Any steroids administered as part of this therapy must be completed ≥3 days prior to the first dose of study medication.
9. Active or history of autoimmune disease that has required systemic treatment within 2 years of the start of study treatment (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).

   Note: Subjects with diabetes type 1, vitiligo, psoriasis, and hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
10. Allogeneic tissue/solid organ transplant, except those not requiring immuno-suppressive treatment.
11. Active infection requiring treatment.
12. History of human immunodeficiency virus (HIV) type 1 or 2 antibodies.
13. Known active hepatitis B whose virus load is greater than 500 IU/mL.
14. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥II), or serious uncontrolled cardiac arrhythmia requiring medication.
15. History or current evidence of any condition, therapy, active infections, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
17. Legally incapacitated or has limited legal capacity.
18. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | First 28 days of treatment
  In subjects in dose escalation
Frequency, severity, and duration of treatment-emergent AEs (TEAEs) | Screening through 90 days after last dose
  For all dose groups according to NCI-CTCAE Version 5.0

SECONDARY OUTCOMES:
Maximum observed concentration at steady state (Cmax-ss) | From first dose through 2 year of treatment
  PK profile of AGEN1223 and balstilimab
Minimum observed concentration at steady state (Cmin-ss) | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
Area under the plasma/serum concentration-time curve within time span t1 to t2 at steady-state (AUC(t1-t2)-ss) | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
Area under the plasma/serum concentration-time curve from time zero to time t (AUC(0-t)) | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
Area under the plasma/serum concentration-time curve from time zero to infinity (AUC(0-∞)) | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
Time to maximum observed concentration (tmax) | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
terminal disposition rate constant (λz) | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
Terminal elimination half-life (t1/2) | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
Systemic clearance (CL) | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
Volume of distribution (Vd). | From first dose through 2 year of treatment
  PK Profile of AGEN1223 and balstilimab
Immunogenicity | From first dose through 2 year of treatment
  Incidence of anti-AGEN1223 antibodies and anti-Balstilimab antibodies
Overall Response Rate | Screening up to 2 years of treatment
  Per RECIST 1.1 based on Investigator assessment
Duration of Response | Screening up to 2 years of treatment
  Per RECIST 1.1 based on Investigator assessment
Disease Control Rate | Screening up to 2 years of treatment
  Including complete and partial responders and stable disease (SD) for at least 12 weeks, per RECIST 1.1 based on Investigator assessment.
Progression-free Survival median and/or rate | Screening up to 2 years of treatment
  As defined in the Statistical Analysis Plan

OTHER OUTCOMES:
PK parameter correlation to pharmacodynamic assessments | Screening up to 1 year of treatment
  Immune cell subpopulations in blood
Characterization of genetic polymorphism of FcyR | Screening up to 2 years of treatment
  In subjects treated with AGEN1223 as single-agent and in combination with balstilimab
Biomarkers of pharmacologic activity | Screening up to 1 year of treatment
  Correlation with tumor responses to AGEN1223 and balstilimab treatment
Biomarkers in tumor tissue and blood | Screening up to 1 year of treatment
  Correlation with tumor responses to AGEN1223 and balstilimab treatment
Median and/or rate of Overall Survival | Up to 12 months after last dose
  As defined in the Statistical Analysis Plan

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agenus Inc.
Locations (4):
- United States (4):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - University of Miami/Sylvester Comprehensive Cancer Center, Miami, Florida
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No